CLINICAL TRIAL: NCT02238249
Title: Post Marketing Surveillance of Alesion® (Epinastine Hydrochloride) Dry Syrup -Special Drug Use-Results Survey of Alesion® Dry Syrup-
Brief Title: Study to Investigate the Safety and Efficacy of Alesion® in Japanese Paediatric Patients With Urticaria
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 262.294
Record Dates: First submitted 2014-09-11; First posted 2014-09-12 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Urticaria
MeSH Terms: conditions — Urticaria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- paediatric patients with urticaria
  Interventions: Drug: Alesion®

INTERVENTIONS:
Drug: Alesion® — Dry Syrup

SUMMARY:
Study to investigate the safety and efficacy of Alesion® Dry Syrup under the proper use in daily clinical practice in Japanese paediatric patients with urticaria

ELIGIBILITY:
Inclusion Criteria:

* All the patients who:

  * haven't treatment experience of epinastine product entered the survey;
  * have urticaria

Exclusion Criteria:

* Alesion® Dry Syrup is contraindicated for the patients with history of hypersensitivity to any ingredients of Alesion® Dry Syrup in package insert. However, it was unknown whether a patient is hypersensitive to the ingredients of the product in almost cases. And this survey was drug utilization study to observe actual use in any patients. Therefore exclusion criteria are not set in the protocol

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with urticaria and without experience in treatment with epinastine are selected by physicians at medical institutions
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2005-10; Primary Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse drug reactions | up to 2 years
  classified by Medical Dictionary for Regulatory Activities (MedDRA)
Incidence of adverse drug reactions classified by patient's background/treatment factors | up to 2 years

SECONDARY OUTCOMES:
Overall assessment of efficacy by investigator on a 3-point scale | after 1 week